CLINICAL TRIAL: NCT06033716
Title: Exploring the Developmental Changes and Relationship Between Resilience and Anxiety and Depression in Elderly Gastric Cancer Survivors: Based on Latent Growth Modeling and Cross-lagged Modeling
Brief Title: Development and Relationship Between Resilience and Anxiety and Depression in Elderly Gastric Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yinning Guo, Principal Investigator, Nanjing Medical University
Other Study IDs: 2020-273-1
Record Dates: First submitted 2023-08-26; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Resilience; Anxiety; Depression
Keywords: gastric cancer; resilience; anxiety; depression; trajectory
MeSH Terms: conditions — Anxiety Disorders; Depression; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement correlation variable — resilience and anxiety and depression

SUMMARY:
This study will explore the dynamic interaction between mental resilience, anxiety and depression in elderly patients with gastric cancer 1 year after surgery, in order to better understand the role of these two factors in patients' mental health, and provide accurate insights for clinical practice and targeted psychological support strategies.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with gastric cancer by endoscopy or pathology
* age ≥60 years old
* radical gastrectomy was proposed
* be able to communicate simply in writing and verbal

Exclusion Criteria:

* received preoperative radiotherapy or chemotherapy;
* combined with other sites of malignant tumors;
* combined with severe heart, liver, lung and renal insufficiency;
* recent using hormones, immunosuppressants;
* with physical disabilities.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: select elderly gastric cancer patients who had undergone cancer surgery and were receiving medical treatment at a tertiary hospital
Sampling Method: Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
resilience | immediately after surgery (T1), three month post-surgery (T2), six months post-surgery (T3), 12 months post-surgery (T4)
  The Chinese version of 10-item Connor-Davidson Resilience Scale (CD-RISC-10), translated and revised by Chinese scholars, was used in this study. Cronbach's alpha for the Chinese version was 0.855, indicating good internal consistency. It was also applied to cancer patients in China. Each of which was scored on a 5-point Likert scale, ranging from 1 to 5 points, from "Never" to "Almost always", with higher scores representing a higher level of psychological resilience.
anxiety | immediately after surgery (T1), three month post-surgery (T2), six months post-surgery (T3), 12 months post-surgery (T4)
  Chinese version of the Hospital Anxiety and Depression Scale (HADS) was used in this study to assess the anxiety and depression of elderly cancer patients, which was developed by Zigmond AS et al. The scale consists of 14 items, including anxiety and depression subscales. Each item is rated on a 4 point scale, and the scores of the anxiety and depression scales range from 0 to 21 points. The Cronbach's α coefficient of the HADS for this study was 0.85.
depression | immediately after surgery (T1), three month post-surgery (T2), six months post-surgery (T3), 12 months post-surgery (T4)
  Chinese version of the Hospital Anxiety and Depression Scale (HADS) was used in this study to assess the anxiety and depression of elderly cancer patients, which was developed by Zigmond AS et al. The scale consists of 14 items, including anxiety and depression subscales. Each item is rated on a 4 point scale, and the scores of the anxiety and depression scales range from 0 to 21 points. The Cronbach's α coefficient of the HADS for this study was 0.85.

CONTACTS AND LOCATIONS:
Locations (1):
- Yinning Guo, Nanjing, Jiangsu, China